CLINICAL TRIAL: NCT04344106
Title: Prone Positioning in Spontaneously Breathing Nonintubated Covid-19 Patient: a Pilot Study (ProCov)
Brief Title: Prone Positioning in Spontaneously Breathing Nonintubated Covid-19 Patient: a Pilot Study
Acronym: ProCov
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ELHARRAR Xavier (Other)
Responsible Party: Sponsor-Investigator, ELHARRAR Xavier, pulmologist, Centre Hospitalier Intercommunal Aix-Pertuis
Organization: Centre Hospitalier Intercommunal Aix-Pertuis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20202703-2
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus Infection; Oxygen Deficiency
MeSH Terms: conditions — Coronavirus Infections; Hypoxia | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prone positioning (Experimental): Participants are all turned to prone position for an optimal minimum duration of 3 hours .
  Tolerance, oxygen saturation, heart rate and position are monitoring during all procedure. Arterial blood gases are realized before, 1 to 2 hours after the beginning of the prone position, and 6 to 12 hours after resupination.
  Interventions: Procedure: Prone positioning

INTERVENTIONS:
Procedure: Prone positioning — The prone positioning consists of placing the patient on his or her stomach with the head on the side, during sessions lasting several hours a day.

SUMMARY:
The prone position consists of placing the patient on his or her stomach with the head on the side, during sessions lasting several hours a day and could help spontaneous ventilate the patient.

DETAILED DESCRIPTION:
SARS-CoV-2 is an RNA virus whose tropism for the respiratory system is responsible for many cases of acute respiratory failure. This can lead to acute respiratory distress syndrome (ARDS) requiring orotracheal intubation and mechanical ventilation. The prone position is a validated intensive care technique in the treatment of ARDS in mechanically ventilated patients. Performing prone position sessions improves patient oxygenation by optimizing the ventilation/perfusion ratios of the posterior areas of the lungs.

There is limited data in the literature on the ventral decubitus in spontaneous ventilation. They are mainly case series or retrospective studies. In the case of the SARS-CoV-2 epidemic, we are seeing patients with posterior lung involvement who may benefit from prone position sessions prior to mechanical ventilation. This maneuver, usually done in an intubated-ventilated-curarized patient, will be done in our spontaneous ventilation study in a conscious patient.The patient will then be placed in prone position with the help of physiotherapists so that the patient is correctly positioned.

The maneuver and the clinical monitoring of the patient's tolerance to the prone position will be done under medical and paramedical supervision, including monitoring of saturation during and after the procedure. A polygraph will also be installed on the patient in order to monitor the patient's position (on the back vs. on the stomach), saturation and heart rate during the entire prone position session. An arterial gasometry will be performed before the patient is placed in the prone position, one hour after and after returning to the supine position.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged at least 18 years;
* Hospitalized in a COVID unit or intensive care unit;
* Spontaneously breathing and with oxygen therapy with nasal canula, mask or High Flow Oxygen Therapy;
* Requiring oxygen therapy ≥ 1l for Sat ≥ 90%;
* COVID 19 positive in RT-PCR or diagnosis on clinicals symptoms and highly evocatives scannographics lesions in an epidemic period;
* Chest scanner without injection within 72 hours prior to inclusion;
* Bilateral scannographic lesions, including posterior condensations and/or posterior predominance of lesions;
* Patient benefiting from French social security, under any regime

Exclusion Criteria:

* acute respiratory distress (polypnea >25 or use of accessory respiratory muscles);
* Alteration of consciousness;
* Active or recent hemoptysis (<1 month);
* Recent Thrombo-Embolic Venous Disease (< 1 month);
* Pericardial effusion;
* Pleural effusion of high abundance, clinical or scannographic;
* Chronic back or cervical pain/ history of spinal surgery/ bone metastases;
* Wounds, facial trauma, tracheal, sternal or facial surgery < 15 days;
* Recent abdominal surgery (< 1 month);
* Intracranial HyperTension > 30mmHg;
* Patient deprived of liberty, under guardianship or curatorship;
* Pregnant or lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of "responder" patients to prone position | 1 hour
  PaO2 improvement of more than 20% after one hour in prone position in spontaneously breathing non intubated COVID-19 patients.

SECONDARY OUTCOMES:
proportion of "persistent responders" patients after prone position | 1 day
  PaO2 improvement of more than 20% at 6 to 12 hours from return to supine position.
Evolution of PaO2 | 1 day
  PaO2 at 1 hour from the start of prone position and at 6 to 12 hours afterreturn to supine position.
Duration of prone positioning and PaO2 evolution | 2 days
  Look for an association between the time spent in Prone positione and persistent responder or not;
Evolution of Spo2 | 1 hour
  proportion of patients improving their arterial saturation within 1 hour of Prone Position
EVA Dyspnea | 1 day
  evolution of the EVA scores for dyspnea at 1 hour from the start of the Prone Position and at 6 hours after the end of the Prone Position
Intolerance to prone positioning | 1 day
  proportion of patients intolerant to prone position (Prone Position <1h);
Tolerance to prone positioning | 1 day
  proportion of patients who can maintain prone position for more than 3 h.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier ELHARRAR, MD, Principal Investigator — Centre Hospitalier Intercommunal Aix-Pertuis (CHIAP), France; Youssef Trigui, MD, Study Director — Centre Hospitalier Intercommunal Aix-Pertuis (CHIAP), France; Stephanie Martinez, MD, Study Chair — Centre Hospitalier Intercommunal Aix-Pertuis (CHIAP), France; Laurence Maulin, MD, Study Chair — Centre Hospitalier Intercommunal Aix-Pertuis (CHIAP), France; Marie Bernardi, MD, Study Chair — Centre Hospitalier Intercommunal Aix-Pertuis (CHIAP), France; Laurent Lefebvre, MD, Study Chair — Centre Hospitalier Intercommunal Aix-Pertuis (CHIAP), France; Thibaut Helbert, MD, Study Chair — Centre Hospitalier Intercommunal Aix-Pertuis (CHIAP), France; Camille begne, MD, Study Chair — Centre Hospitalier Intercommunal Aix-Pertuis (CHIAP), France
Locations (1):
- CHI Aix-Pertuis, Aix-en-Provence, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun Q, Qiu H, Huang M, Yang Y. Lower mortality of COVID-19 by early recognition and intervention: experience from Jiangsu Province. Ann Intensive Care. 2020 Mar 18;10(1):33. doi: 10.1186/s13613-020-00650-2. No abstract available. PMID 32189136
- [Background] Scaravilli V, Grasselli G, Castagna L, Zanella A, Isgro S, Lucchini A, Patroniti N, Bellani G, Pesenti A. Prone positioning improves oxygenation in spontaneously breathing nonintubated patients with hypoxemic acute respiratory failure: A retrospective study. J Crit Care. 2015 Dec;30(6):1390-4. doi: 10.1016/j.jcrc.2015.07.008. Epub 2015 Jul 16. PMID 26271685
- [Background] Ding L, Wang L, Ma W, He H. Efficacy and safety of early prone positioning combined with HFNC or NIV in moderate to severe ARDS: a multi-center prospective cohort study. Crit Care. 2020 Jan 30;24(1):28. doi: 10.1186/s13054-020-2738-5. PMID 32000806
- [Background] Munshi L, Del Sorbo L, Adhikari NKJ, Hodgson CL, Wunsch H, Meade MO, Uleryk E, Mancebo J, Pesenti A, Ranieri VM, Fan E. Prone Position for Acute Respiratory Distress Syndrome. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2017 Oct;14(Supplement_4):S280-S288. doi: 10.1513/AnnalsATS.201704-343OT. PMID 29068269
- [Background] Gattinoni L, Taccone P, Carlesso E, Marini JJ. Prone position in acute respiratory distress syndrome. Rationale, indications, and limits. Am J Respir Crit Care Med. 2013 Dec 1;188(11):1286-93. doi: 10.1164/rccm.201308-1532CI. PMID 24134414
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Shi H, Han X, Jiang N, Cao Y, Alwalid O, Gu J, Fan Y, Zheng C. Radiological findings from 81 patients with COVID-19 pneumonia in Wuhan, China: a descriptive study. Lancet Infect Dis. 2020 Apr;20(4):425-434. doi: 10.1016/S1473-3099(20)30086-4. Epub 2020 Feb 24. PMID 32105637